CLINICAL TRIAL: NCT01600872
Title: Oxidative Stress and BPA Impact With PCOS
Brief Title: Oxidative Stress and Bisphenol A (BPA) Impact With Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ming-I Hsu (Other)
Responsible Party: Sponsor-Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Organization: Taipei Medical University WanFang Hospital (Other)
Other Study IDs: WFH-TMU-PCOS-201112030
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Oxidative Stress; Endocrine Disrupting Chemicals; Polycystic Ovary Syndrome
Keywords: EDCs; PCOS; TAS; TOS; ROS; Oxidative Stress, Endocrine-Disrupting Chemicals, Polycystic Ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gruop 1
- Group 2

SUMMARY:
Both oxidative stress and Bisphenol A (BPA) had been associated with polycystic ovary syndrome (PCOS). BPA, one of endocrine-disrupting chemicals (EDCs), is an environmental estrogen used in the synthesis of plastics, is a "high-volume production" chemical with widespread human exposure. BPA was been reported in several female reproductive disturbance. However, the pathological pathway of BPA impact on female reproductive system had not been well-understood. Reactive oxygen species (ROS) have a role in the modulation of gamete quality and gamete interaction. Persistent and elevated generation of ROS leads to a disturbance of redox potential that in turn causes oxidative stress (OS). The first part of The investigators study is aim to evaluate the oxidative stress impact on the biochemical parameters in women with PCOS; the secondary part of the investigators study is to investigate the BPA on the clinical and biochemical of women with PCOS; finally, the investigators plan to test the hypothesis that BPA might increase oxidative stress and then elevated ROS in women with menstrual disturbance, furthermore, the role of oxidative stress and BPA impact on insulin resistance and metabolic disturbance will be also investigated.

Study and control cases will be included. Serum total oxidant status (TOS), total antioxidant status (TAS), Bisphenol A (BPA), and clinical/biochemical parameters will be obtained for all cases. Oxidative stress and BPA will be evaluated with all clinical/biochemical parameters for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Normal health control
2. Women with reproductive endocrine disturbance menstrual irregularity, and/or polycystic ovary syndrome.

Exclusion Criteria:

* The following subjects were excluded from the study and control populations:

  1. women who experienced menarche less than 3 years prior to the start of the study;
  2. women who received hormones, antioxidants or drugs for major medical diseases such as diabetes or cardiovascular disease; and
  3. women who were older than 45.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal health control and Women with reproductive endocrine disturbance menstrual irregularity, and/or polycystic ovary syndrome.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan